CLINICAL TRIAL: NCT05553262
Title: A Three-years Project for Assistance and Dental Care of Children With Autistic Spectrum Disorder at the Community Dentistry Unit - Piove di Sacco Hospital (Padua, Italy)
Brief Title: A Protocol to Streamline Dental Care in Autistic Children
Acronym: DentAutism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Collaborators: Azienda Ulss 6 Euganea (Other); Nastrificio Victor S.p.A. (Unknown)
Responsible Party: Principal Investigator, MUCIGNAT CARLA, Principal Investigator, University of Padova
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUTISM
Record Dates: First submitted 2022-09-14; First posted 2022-09-23 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; Dentistry
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Behavior Therapy

STUDY DESIGN:
Intervention Model Description: Both treated and control groups will receive the same clinical intervention (dental care) when needed. Treated group will have visits every two months, visual pedagogy and caregiver instructions for oral hygiene maintenance at home. Control group will receive dentist visits twice a year (or more often if clinically required) according to Italian Ministry of Health guidelines for pediatric dentistry.
Masking Description: No masking is possible because caregivers must accept and comply a strict schedule of visits for three years. The dentists are aware of the participation to the protocol because they use additional supports and strategies, like a longer duration of the visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral support (Experimental): Usual clinical intervention and in addition: visual pedagogy, instruction of caregivers, a visit every two months for three years, fixed duration of the visit (one hour) regardless of patients' collaboration. General anesthesia if needed.
  Interventions: Behavioral: Behavioral support
- Control No behavioral support (No Intervention): Usual clinical treatment (dentist visit and treatments). No visual pedagogy and instruction of caregivers. Twice a year schedule (more if needed), duration of the visits according to compliance. General anesthesia if needed.

INTERVENTIONS:
Behavioral: Behavioral support — Behavioral support as described under 'Arm description'.
  Arms: Behavioral support

SUMMARY:
The investigators aim at creating a dedicated pathway to allow accessibility to dental care for ASD children within a hospital Dentistry Department, in order to diminish the need for general anesthesia. Visual pedagogy, parent training, a strict schedule for appointments (every two months) spanning over three years and longer duration of dedicated examination are set up for a group of ASD children, whose behavior is compared to that of children seen one or twice a year.

DETAILED DESCRIPTION:
Treated group:

Enrollment: caregivers receive instructions and a visual pedagogy aid with instructions for toothbrushing. They complete also enrollment and informed consent forms.

At the first visit: caregivers receive a dental mirror to be used at home. Children are free to explore the office and dental room.

Subsequent visits, every two months for three years: trials are made to establish contact with children, make them seat at the dentist's chair, execute dental visits and treatments as needed.

Control group: subjects (similar inclusion and exclusion criteria) that access the Department for clinical reasons or control visits, but cannot comply with the strict two-months schedule.

ELIGIBILITY:
Inclusion Criteria:

* Age: 4 to 13 years old at the beginning of the treatment,
* Diagnosis: formally diagnosed by a Neuro-psychiatrist and recognized by authorities (for school support) as having Autistic Spectrum Disorder (ASD), possibly also in the frame of genetic syndromes, or Pervasive Developmental Disorder-Not Otherwise Specified (PDD-NOS), a diagnosis present in DSM 4 and merged to ASD in DSM 5.

Exclusion Criteria:

* Age outside the selected range
* additional diseases, preventing autonomous oral hygiene (e.g., motor diseases),
* for the Treated Group: familiarity with dental treatments (possible one or few visits in the past, but not on a regular base)

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 170 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Collaboration | Change in degree of collaboration from baseline at 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 34, 36 months.
  Degree of collaboration on Frankl's scale, from 0 (none) to 3 (optimal)

SECONDARY OUTCOMES:
Acceptance | Year 1, month 2
  Acceptance of every action or instrument: Yes/No
Acceptance | Year 1, month 4
  Acceptance of every action or instrument: Yes/No
Acceptance | Year 1, month 6
  Acceptance of every action or instrument: Yes/No
Acceptance | Year 1, month 8
  Acceptance of every action or instrument: Yes/No
Acceptance | Year 1, month 10
  Acceptance of every action or instrument: Yes/No
Acceptance | Year 1, month 12
  Acceptance of every action or instrument: Yes/No
Acceptance | Year 2, month 2
  Acceptance of every action or instrument: Yes/No
Acceptance | Year 2, month 4
  Acceptance of every action or instrument: Yes/No
Acceptance | Year 2, month 6
  Acceptance of every action or instrument: Yes/No
Acceptance | Year 2, month 8
  Acceptance of every action or instrument: Yes/No
Acceptance | Year 2, month 10
  Acceptance of every action or instrument: Yes/No
Acceptance | Year 2, month 12
  Acceptance of every action or instrument: Yes/No
Acceptance | Year 3, month 2
  Acceptance of every action or instrument: Yes/No
Acceptance | Year 3, month 4
  Acceptance of every action or instrument: Yes/No
Acceptance | Year 3, month 6
  Acceptance of every action or instrument: Yes/No
Acceptance | Year 3, month 8
  Acceptance of every action or instrument: Yes/No
Acceptance | Year 3, month 10
  Acceptance of every action or instrument: Yes/No
Acceptance | Year 3, month 12
  Acceptance of every action or instrument: Yes/No

CONTACTS AND LOCATIONS:
Overall Officials: Carla Mucignat, Ph.D., Principal Investigator — University of Padova
Locations (1):
- Piove di Sacco Hospital, Piove di Sacco, PD, Italy

IPD SHARING:
Plan to Share IPD: No
Only anonymized data, including age, sex, diagnosis and the collected measurements, will be made available to other researchers. Individual Participant data that allow identification of the single participant cannot be shared, as requested by the Ethical Committee.

REFERENCES:
- [Background] AlBhaisi IN, Kumar MSTS, Engapuram A, Shafiei Z, Zakaria ASI, Mohd-Said S, McGrath C. Effectiveness of psychological techniques in dental management for children with autism spectrum disorder: a systematic literature review. BMC Oral Health. 2022 May 6;22(1):162. doi: 10.1186/s12903-022-02200-7. PMID 35524299
- [Background] Aljubour A, AbdElBaki M, El Meligy O, Al Jabri B, Sabbagh H. Effect of Culturally Adapted Dental Visual Aids on Oral Hygiene Status during Dental Visits in Children with Autism Spectrum Disorder: A Randomized Clinical Trial. Children (Basel). 2022 May 5;9(5):666. doi: 10.3390/children9050666. PMID 35626843
- [Background] Alvares GA, Mekertichian K, Rose F, Vidler S, Whitehouse AJO. Dental care experiences and clinical phenotypes in children on the autism spectrum. Spec Care Dentist. 2023 Jan;43(1):17-28. doi: 10.1111/scd.12746. Epub 2022 Jun 2. PMID 35654391
- [Background] Shalabi MASA, Khattab NMA, Elheeny AAH. Picture Examination Communication System Versus Video Modelling in Improving Oral Hygiene of Children with Autism Spectrum Disorder: A Prospective Randomized Clinical Trial. Pediatr Dent. 2022 Jan 15;44(1):25-31. PMID 35232533
- [Background] Yost Q, Nelson T, Sheller B, McKinney CM, Tressel W, Chim AN. Children with Autism Spectrum Disorder Are Able to Maintain Dental Skills: A Two-Year Case Review of Desensitization Treatment. Pediatr Dent. 2019 Sep 15;41(5):397-403. PMID 31648672